CLINICAL TRIAL: NCT04150588
Title: The Correlation Between Müller's Muscle-Conjunctival Resection and Phenylephrine Test
Brief Title: The Correlation Between MMCR and Phenylephrine Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Sheba-19-6248-PA-CTIL
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: the Correlation Between Erin Test and Müller's Muscle-Conjunctival Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good reaction to Efrin test
  Interventions: Drug: Efrin drops
- Unsatisfied reaction to Efrin test
  Interventions: Drug: Efrin drops

INTERVENTIONS:
Drug: Efrin drops — The amount that the eyelid rise after Erin drops before surgery

SUMMARY:
The propose of the study is the examine the association between the amount that the eyelid rise 3 months after surgery and the reaction to Efrin test before surgery

ELIGIBILITY:
Inclusion Criteria:

* patients with ptosis
* patients that react to Efrin test

Exclusion Criteria:

* Other eye diseases
* other eye surgeries

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ptosis over 18 YO that react to efrin test
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
The reaction to efrin test before surgery | 15 minutes

SECONDARY OUTCOMES:
The amount that the eyelid rise after surgery | 3 MONTHS postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided